CLINICAL TRIAL: NCT06350552
Title: Investigating the Prevalence of Hyper Kyphosis and Forward Head Posture in Dialysis Patients
Brief Title: Prevalence of Postural Abnormalities in Dialysis Patients
Status: Completed | Type: Observational
Sponsor: Pardis Specialized Wellness Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PA224ES-1-03
Record Dates: First submitted 2024-03-19; First posted 2024-04-05 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: End Stage Renal Disease; Hemodialysis Complication; Peritoneal Dialysis Complication
Keywords: Postural Kyphosis; Postural, Thoracic Kyphosis; Physical Function; Fall; Balance
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Hemodialysis: They will be assessed for postural abnormalities. Also, they will do some physical function tests.
- Peritoneal Dialysis: They will be assessed for postural abnormalities. Also, they will do some physical function tests.

SUMMARY:
The goal of this observational study is to investigate and compare the prevalence of forward head , hyper kyphosis and balance in hemodialysis and peritoneal dialysis patients. The main questions it mains to answer are:

What is the prevalence of forward head posture in hemodialysis and peritoneal dialysis patients? What is the prevalence of hyper kyphosis in hemodialysis and peritoneal dialysis patients? Is there any relation between postural abnormalities and physical function in hemodialysis and peritoneal dialysis patients?

Participants will answer 2 questionnaires and will do some functional tests.

DETAILED DESCRIPTION:
Given the global rise in fall rates and associated medical costs in the past decade, it is crucial to identify factors that contribute to fall risk in order to mitigate the occurrence of falls and reduce their adverse consequences.

One significant factor that increases the likelihood of falls is the presence of a balance disorder. The Forward head posture (FHP) can adversely affect one's static balance. FHP characterized by the bending forward of the lower cervical spine and the bending backward of the upper cervical spine. The prevalence of FHP rises as one gets older and has been associated with an elevated risk of falls, altered limits of stability, and changes in the musculoskeletal structures of the cervical spine. FHP can significantly impact respiratory function by weakening the muscles involved in breathing.

Alterations in the positioning of the center of gravity can have a detrimental impact on the control of body balance . Balance can also be affected by thoracic hyper kyphosis, which refers to an excessive curvature of the thoracic spine. When compensation in the lumbar spine and hip region is insufficient, hyper kyphosis may shift the body's center of mass forward, leading to gait disorders and disrupted balance.

Changes in posture, like thoracic hyper kyphosis and loss of lumbar lordosis arch seem to contribute to the increased postural instability and leading to a greater likelihood of falls among older adults living in the community. Hyper kyphosis may act as an indicator of an elevated risk of falls. Internationally, thoracic hyper kyphosis has a high prevalence, and studies have shown that it is associated with impaired performance in balance, gait, and cardiopulmonary function tests among older adults.

The likelihood of hyper kyphosis and FHP, followed by increased falls in elderly individuals and women, is attributed to factors such as reduced physical activity, lower bone density, weaker muscles, and decreased overall body strength . Considering the presence of these conditions in dialysis patients, it is likely that these patients are also at an increased risk of kyphosis and FHP, and consequently, they face the risk of falls.

The study of postural abnormalities in patients undergoing hemodialysis (HD) and peritoneal dialysis (PD) makes it possible to identify prevention and safety promotion strategies for individuals with chronic kidney disease. Thus, the objectives of this study are to identify the prevalence of forward head and hyper kyphosis as well as their adverse outcomes in people with chronic kidney disease undergoing two dialysis modalities.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria will be as follows:

1. age ≥18 years;
2. on dialysis for ≥3 months;
3. able to walk without assistance (walking device such as cane or walker allowed); and
4. ability to provide informed consent and complete the questionnaires.

Exclusion Criteria:

The exclusion criteria will include

1. diagnosis of mental or cognitive disorders;
2. unstable conditions; and
3. hospitalization in the previous 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis and peritoneal dialysis patients being treated with the same respective dialysis modalities for at least 3 months and being ambulatory (with or without assistive device) will be included.
  But non-ambulatory patients having significant cognitive dysfunction, progressive degenerative,neurologic disease or severe rheumatologic or orthopedic conditions, angina upon exertion, or myocardial infarction or cardiac surgery within the last year will be excluded.
Sampling Method: Probability Sample
Enrollment: 395 (Actual)
Dates: Start 2024-04-28 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of thoracic hyper kyphosis | Through out study completion, an average of 1 weeks
  Thoracic hyper kyphosis using the flexicurve approach, the procedure will involve utilizing a 60 cm flexible ruler (Trident®), millimeter paper, adhesive tape, pen, and a specific formula will be documented in Microsoft Excel.
Prevalence of forward head | Through out study completion, an average of 1 weeks
  The digital imaging technique (knee registry application) will be utilized to assess head and neck posture in a standing position. A mobile device will be positioned 150 cm away on a tripod stand, adjusting the height to align with the subject's shoulder level. The subject will be directed to face the camera straight on and then to the side. A photo will be captured and saved in jpg format using the knee registry application. A line will be drawn from the spinous process to the tragus of the ear, and the angle will subsequently be measured. The craniovertebral angle will often be employed as a diagnostic tool for identifying forward head.

SECONDARY OUTCOMES:
Balance level | Through out study completion, an average of 1 weeks
  Timed Up & Go Test (TUG) will be used for balance evaluation. During this test, participants will be required to stand up from a chair, walk a distance of 3 meters, turn around, walk back to the chair, and sit down while the researchers will record the time taken for the entire process. A shorter time taken in this test will be indicative of better dynamic balance. Generally, if a participant completes the test within 10 seconds, it will be considered as having a normal dynamic balance
Cardiopulmonary function's level | Through out study completion, an average of 1 weeks
  The 6-minute walk test (6MWT) will be frequently utilized as one of the most common walk tests and will be used to assess cardiopulmonary function. The 6MWT will take place on a level, 30-meter-long square within the local community. Participants will be instructed to walk for six minutes to cover as much distance as they can. Prior to the test, the participants' blood pressure and heart rate will be recorded. The researcher will measure the distance walked. An outcome of ≥375 meters suggests that cardiopulmonary function is either near normal or normal, whereas a result of <375 meters suggests impaired cardiopulmonary function
Fall risk level | Through out study completion, an average of 1 weeks
  Tinetti (ICC > 0.8) Will be used to examine gait dysfunctions and static balance. Patients scoring less than 11 on 12 on the Tinetti test are considered being at an increased risk of falls. The test comprises two short sections that contain one examining static balance abilities in a chair and then standing, and the other gait.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Ali Tabibi, Dr, Principal Investigator — Pardis Specialized Wellness Institute; Bobby Cheema, Dr, Study Director — School of Health Sciences, Western Sydney University, Campbelltow, NSW 2560, Australia
Locations (1):
- Khorshid Dialysis Center, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the published article, after deidentification are to be shared.
Supporting Information: Study Protocol
Time Frame: The data will be available after the paper is published. No end date.
Access Criteria: Data will be accessible with no criteria. Anyone who wishes will have access to data.

REFERENCES:
- [Result] Rossier A, Pruijm M, Hannane D, Burnier M, Teta D. Incidence, complications and risk factors for severe falls in patients on maintenance haemodialysis. Nephrol Dial Transplant. 2012 Jan;27(1):352-7. doi: 10.1093/ndt/gfr326. Epub 2011 Jun 7. PMID 21652549
- [Result] Wang HH, Wu JL, Lee YC, Ho LC, Chang MY, Liou HH, Hung SY. Risk of Serious Falls Between Hemodialysis and Peritoneal Dialysis Patients: A Nationwide Population-based Cohort Study. Sci Rep. 2020 May 8;10(1):7799. doi: 10.1038/s41598-020-64698-7. PMID 32385311
- [Result] Muir SW, Berg K, Chesworth B, Klar N, Speechley M. Quantifying the magnitude of risk for balance impairment on falls in community-dwelling older adults: a systematic review and meta-analysis. J Clin Epidemiol. 2010 Apr;63(4):389-406. doi: 10.1016/j.jclinepi.2009.06.010. Epub 2009 Sep 9. PMID 19744824
- [Result] Kado DM, Huang MH, Karlamangla AS, Barrett-Connor E, Greendale GA. Hyperkyphotic posture predicts mortality in older community-dwelling men and women: a prospective study. J Am Geriatr Soc. 2004 Oct;52(10):1662-7. doi: 10.1111/j.1532-5415.2004.52458.x. PMID 15450042
- [Result] Li WY, Chau PH, Dai Y, Tiwari AF. The Prevalence and Negative Effects of Thoracic Hyperkyphosis on Chinese Community-Dwelling Older Adults in Wuhan, Hubei Province, China. J Nutr Health Aging. 2021;25(1):57-63. doi: 10.1007/s12603-020-1441-1. PMID 33367463
- [Result] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Result] Buracchio T, Dodge HH, Howieson D, Wasserman D, Kaye J. The trajectory of gait speed preceding mild cognitive impairment. Arch Neurol. 2010 Aug;67(8):980-6. doi: 10.1001/archneurol.2010.159. PMID 20697049
- [Result] Padilla J, Krasnoff J, Da Silva M, Hsu CY, Frassetto L, Johansen KL, Painter P. Physical functioning in patients with chronic kidney disease. J Nephrol. 2008 Jul-Aug;21(4):550-9. PMID 18651545